CLINICAL TRIAL: NCT06958263
Title: Factors Associated With Sensitization in Patients With Chronic Low Back Pain
Brief Title: Relationship Between Low Back Pain and Sensitization
Status: Recruiting | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Musa Güneş, Principal Investigator, PhD, Karabuk University
Other Study IDs: Karabuk-003
Record Dates: First submitted 2025-04-25; First posted 2025-05-06 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Higher sensitization: Patients with chronic non-specific low back pain with high sensitization will be included.
- Normal sensitization: Patients with chronic non-specific low back pain with normal sensitization will be included.

SUMMARY:
Chronic non-specific low back pain is a common health problem that significantly affects the quality of life of individuals. Increased pain intensity leads to deficiencies in the body's sensory organization, resulting in decreased awareness. This can lead to dysfunction in body awareness, which is known as the ability of individuals to perceive the sensations and conditions of their bodies. Body awareness plays a critical role in pain management and mobility. Chronic pain causes constant stimulation in the nervous system, causing central sensitization, which is when the central nervous system becomes overly sensitive to pain signals. As a result, a decrease in the pain threshold, constant pain, and increased muscle tension occur. Increased pain intensity and decreased awareness can result in a decrease in the maintenance of optimal functions, affecting muscular endurance. Inadequate muscular endurance can increase low back pain and make it difficult for individuals to perform their daily activities. Therefore, this study aims to examine the relationship between body awareness, central sensitization, disability, and muscular endurance in patients with chronic non-specific low back pain.

DETAILED DESCRIPTION:
Body awareness plays a critical role in pain management and mobility. Individuals with high body awareness can better manage their pain, which can contribute to a decrease in disability levels. Chronic pain causes constant stimulation in the nervous system, which causes central sensitization, which is when the central nervous system becomes oversensitive to pain signals. As a result, a decrease in the pain threshold, constant pain, and increased muscle tension occur. In addition, central sensitization can cause the body to be more vulnerable to injuries due to the body being in an overstimulated state. Increased pain intensity and decreased awareness can result in a decrease in the maintenance of optimal functions, affecting muscular endurance. Inadequate muscular endurance can increase low back pain and make it difficult for individuals to perform their daily activities. The literature has attempted to emphasize the relationship between pain, disability, and body awareness in various populations. However, the relationship between body awareness and central sensitization has not been sufficiently studied. Sensitization in the body as a result of central sensitization may be associated with changes in awareness. Understanding these complex relationships is important for developing appropriate treatment strategies in the rehabilitation and clinical follow-up process. Therefore, this study aims to investigate the relationship between body awareness, central sensitization, disability and muscular endurance in patients with chronic non-specific low back pain. Patients with chronic non-specific low back pain will be included in the study. Body awareness, central sensitization, pain intensity, muscular endurance and disability levels of the patients will be evaluated. The data obtained from the study will be analyzed appropriately.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Being diagnosed with chronic non-specific low back pain (Pain between the gluteal folds and the 12th ribs that lasts at least 12 weeks and has no known pathoanatomical cause)
* Being willing to participate in the study

Exclusion Criteria:

* Having a psychological disorder, mental disorder, cancer and severe depression
* Having a history of primary or metastatic spinal malignancy, spinal fracture
* Having a neurological disease (Hemiplegia, Multiple Sclerosis, Parkinson's, etc.)
* Being diagnosed with advanced osteoporosis
* Having a history of surgery or acute infection in the lumbar region

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic non-specific low back pain will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Central sensitization | Baseline
  Central sensitization will be assessed with the "Central Sensitization Scale". The total score range is between 0-100 points. As the score increases, sensitization increases and 40 points and above are considered higher sensitization.
Pain severity | Baseline
  Pain intensity will be assessed with Vizüel Analog Scale (VAS). VAS varies between 0-10 and the higher the score, the greater the pain.
Pain pressure threshold | Baseline
  Pressure pain threshold will be measured with an algometer in kg. High values indicate a high pain threshold.
Disability levels | Baseline
  Disability will be measured by the Oswestry Disability Index. The total score ranges from 0-100 and the higher the score, the higher the level of disability.
Body awereness | Baseline
  It will be measured with a body awareness survey. The total score varies between 18-126 and as the score increases, awareness increases
Low back awereness | Baseline
  It will be measured with the Fremantle Waist Awareness Questionnaire (FBFA). The total score varies between 0-36 and the awareness decreases as the score increases
Trunk muscle endurance | Baseline
  The Stabilizer Pressure Biofeedback Unit will be used to evaluate the multifidus muscle endurance. The time maintained at 40 mmHg pressure will be recorded. As the time increases, the endurance increases.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Güneş, PhD, Study Director — Karabuk University; Seher İmanur, Principal Investigator — Karabuk University; Elif Aydoğan, Principal Investigator — Karabuk University; Bedirhan Turan, Principal Investigator — Karabuk University; Aydın Sinan Apaydın, PhD, Principal Investigator — Karabuk University
Locations (1):
- Karabuk University, Physiotherapy and Rehabilitation Application and Research Center, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nijs J, Van Houdenhove B, Oostendorp RA. Recognition of central sensitization in patients with musculoskeletal pain: Application of pain neurophysiology in manual therapy practice. Man Ther. 2010 Apr;15(2):135-41. doi: 10.1016/j.math.2009.12.001. Epub 2009 Dec 24. PMID 20036180
- [Result] Colgan DD, Eddy A, Green K, Oken B. Adaptive body awareness predicts fewer central sensitization-related symptoms and explains relationship between central sensitization-related symptoms and pain intensity: A cross-sectional study among individuals with chronic pain. Pain Pract. 2022 Feb;22(2):222-232. doi: 10.1111/papr.13083. Epub 2021 Nov 11. PMID 34651401